CLINICAL TRIAL: NCT00299000
Title: A Phase 4 Multi-center, Multi-national, Open-label, Randomized, Two Dose Level Study of Naglazyme(TM) (Galsulfase) in Infants With Maroteaux-Lamy Syndrome (MPS VI)
Brief Title: A Phase 4 Two Dose Level Study of Naglazyme(TM) (Galsulfase) in Infants With MPS VI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Celeste Decker, MD, BioMarin Pharmaceutical Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ASB-008
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Results first posted 2010-10-15 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Mucopolysaccharidosis VI; Maroteaux-Lamy Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis VI | interventions — galsulfase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naglazyme, 1.0 mg/kg (Other): Dose comparison
  Interventions: Drug: Naglazyme
- Naglazyme, 2.0 mg/kg (Other): Dose Comparison
  Interventions: Drug: Naglazyme

INTERVENTIONS:
Drug: Naglazyme — Weekly infusion for minimum of 52 weeks. Naglazyme is diluted in sterile 0.9% sodium chloride solution
  Other Names: recombinant human N-acetylgalactosamine 4-sulfatase; rh-arylsulfatase B; rhASB

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of two dose levels of Naglazyme in infants under the age of one year who have MPS VI by monitoring physical appearance, x-ray of the skeletal system and growth.

DETAILED DESCRIPTION:
The primary objective of the study was to evaluate the efficacy of two dose levels of Naglazyme in preventing the progression of skeletal dysplasia in infants under the age of one year who have MPS VI by monitoring physical appearance, x-ray of the skeletal system and growth.

The secondary objective of the study was to evaluate the efficacy of the two dose levels of Naglazyme in preventing several measures of disease progression in infants under the age of one year who have MPS VI by monitoring urinary GAGs, gross and fine motor function, cardiac function, vision, hearing, and use of health resources.

The safety objective of the study was to evaluate the safety of two dose levels of Naglazyme in infants under the age of one year who have MPS VI.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by a parent or legal guardian
* Parent or legal guardian willing and able to comply with all study procedures
* Equal to or greater than 36 weeks estimated gestational age by physical exam at birth
* Has a diagnosis of MPS VI based on a documented prenatal diagnosis or fibroblast or leukocyte N-acetylgalactosamine 4-sulfatase (ASB) enzyme activity level of less than 10% of the lower limit of the normal range of the measuring laboratory
* Is less than one year of age
* Has no evidence of skeletal dysplasia based on physical exam

Exclusion Criteria:

* Parent of legal guardian perceived to be unreliable or unavailable for study participation
* Use of any investigational drug within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments
* Has concurrent disease or condition that would interfere with study participation or safety (i.e., has previously undergone hematopoietic stem cell transplantation such as bone marrow or cord blood transplantation, or major organ transplantation)
* Any condition that, in the view of the principle investigator, renders the subject at high risk from treatment compliance and/or completing the study
* Has known hypersensitivity to Naglazyme
* Has previously received Naglazyme

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2006-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Decker, MD, Study Director — BioMarin Pharmaceutical
Locations (4):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Oakland, Oakland, California
- Hospital Femme Mere Enfant Centre, Lyon, France
- Hospital PediAtrico de Coimbra, Coimbra, Portugal

REFERENCES:
- [Derived] Garcia P, Phillips D, Johnson J, Martin K, Randolph LM, Rosenfeld H, Harmatz P. Long-term outcomes of patients with mucopolysaccharidosis VI treated with galsulfase enzyme replacement therapy since infancy. Mol Genet Metab. 2021 May;133(1):100-108. doi: 10.1016/j.ymgme.2021.03.006. Epub 2021 Mar 14. PMID 33775523
- [Derived] Harmatz PR, Garcia P, Guffon N, Randolph LM, Shediac R, Braunlin E, Lachman RS, Decker C. Galsulfase (Naglazyme(R)) therapy in infants with mucopolysaccharidosis VI. J Inherit Metab Dis. 2014 Mar;37(2):277-87. doi: 10.1007/s10545-013-9654-7. Epub 2013 Oct 10. PMID 24108527
- See also: BioMarin Pharmaceutical Inc Website — http://www.BRMN.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Global study sites were hospitals.
  First Enrollment: 08MAY2006
  Last Dose: 30APR2009
Groups:
- Naglazyme, 1.0 mg/kg; Naglazyme, 2.0 mg/kg: weekly infusions for minimum of 52 weeks
Period: Overall Study
Arm/Group | Naglazyme, 1.0 mg/kg | Naglazyme, 2.0 mg/kg
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naglazyme, 1.0 mg/kg | Naglazyme, 2.0 mg/kg | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: months] | 6.05 (3.89) | 12.4 (0.42) | 9.23 (4.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-Hispanic | 1 | 1 | 2
  Hispanic/Latino | 1 | 0 | 1
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 0 | 2
  France | 0 | 1 | 1
  Portugal | 0 | 1 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Change in Urinary Glycosaminoglycan Levels
Description: Change in urinary GAG levels was calculated from baseline to week 52 of treatment.
Time Frame: minimum 52 weeks of dosing
Population: Intention to treat.
Measure: Mean (Standard Deviation); unit: ug/mg creatinine
Arm/Group | Naglazyme, 1.0 mg/kg | Naglazyme, 2.0 mg/kg
Number analyzed (Participants) | 2 | 2
ug/mg creatinine
  Baseline | 1041.87 (86.32) | 698.95 (142.34)
  Week 52 | 261.15 (54.38) | 178.10 (42.43)
  Change from Baseline to Week 52 | -780.72 (140.69) | -520.85 (99.91)

2. Primary Outcome: Change in Height
Time Frame: 52 weeks
Population: Intention to treat.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Naglazyme, 1.0 mg/kg | Naglazyme, 2.0 mg/kg
Number analyzed (Participants) | 2 | 2
centimeters
  Height at baseline | 67.3 (5.1) | 80.3 (1.8)
  Height at week 52 | 81.9 (1.8) | 91.3 (5.2)
  Change in height | 14.6 (6.9) | 11.0 (7.0)

3. Primary Outcome: Change in Weight
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Naglazyme, 1.0 mg/kg | Naglazyme, 2.0 mg/kg
Number analyzed (Participants) | 2 | 2
kilograms
  weight at baseline | 7.1 (.3) | 10.2 (.6)
  weight at week 52 | 11.3 (.3) | 13.3 (1.0)
  change in weight | 4.2 (.6) | 3.1 (1.6)

4. Primary Outcome: Change in Haed Circumference
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Naglazyme, 1.0 mg/kg | Naglazyme, 2.0 mg/kg
Number analyzed (Participants) | 2 | 2
centimeter
  head circumference at baseline | 43.5 (3.0) | 49.1 (.5)
  head circumference at 52 weeks | 48.5 (1.0) | 51.8 (.8)
  Change in head circumference | 5.0 (4.0) | 2.7 (1.3)

ADVERSE EVENTS:
Time Frame: All patients received weekly infusions of Nagalzyme for a minimum of 52 weeks. The range in time of exposure to Naglazyme for the duration of the study was 52.9 to 153.30 weeks.
Arm/Group | Naglazyme, 1.0 mg/kg | Naglazyme, 2.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 2/2 | 2/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naglazyme, 1.0 mg/kg (N=2) | Naglazyme, 2.0 mg/kg (N=2)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Cast application (Surgical and medical procedures) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Poor venous access (Vascular disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naglazyme, 1.0 mg/kg (N=2) | Naglazyme, 2.0 mg/kg (N=2)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 2 (3)
Ear infection (Infections and infestations) | 2 (2) | 2 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (15) | 1 (1)
Pyrexia (General disorders) | 2 (8) | 1 (31)
Rhinitis (Infections and infestations) | 1 (3) | 2 (3)
Umbilical hernia (Gastrointestinal disorders) | 2 (3) | 1 (1)
Upper respiratory tract infections (Infections and infestations) | 2 (9) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (3)

LIMITATIONS AND CAVEATS:
Given the small number of patients (4) represented in this study, the outcomes observed in this study may not reflect or predict outcomes observed by physicians in clinical practice.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of the results shall be made by the Sponsor in a joint publication. If such a multicenter publication is not submitted within 12 months after conclusion of the study, the PI may publish the results from site individually, subject however to comply with the other terms of the agreement.